CLINICAL TRIAL: NCT07358117
Title: Viral Infections of the Central Nervous System: Diagnosis and Clinical Outcome
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LCR-VIR
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Infection; Virus Disease; CNS Infection
MeSH Terms: conditions — Infections; Virus Diseases; Central Nervous System Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- immunocompetent adults
- immunocompetent pediatric
- adult and paediatric immunosuppressed

SUMMARY:
Central Nervous System (CNS) infections are caused by bacteria, viruses, fungi, helminths, with several clinical aspects. Studies in the literature generally focus on a single patient type, and no experiences have been reported in which immunosuppressed and immunocompetent adult and pediatric patients were simultaneously examined. Our study will include all possible patient types (immunocompetent adults, immunocompetent pediatric patients, and subjects immunosuppressed by co-softness), to try to more precisely define the clinical and population characteristics of patients who have had an episode of CNS viral infection. These indications may be useful in the future to more specifically guide diagnostic investigations on patients considered at risk.

DETAILED DESCRIPTION:
The objectives are: 1) to verify whether the different categories of patients present a different distribution of etiological agents (Citomegalovirus, Herpes Simplex Virus 1, Herpes Simplex Virus 2, Human Herpesvirus 6, Varicella Zoster Virus, Epstein-Barr Virus, Enterovirus) for CNS infection; 2) to verify whether the course and clinical manifestations of the disease can be associated with the identified etiological agent and the type of patient; 3) to describe the results of instrumental tests (EEC and/or MRI and/or CT) in patients who tested positive for a neurotropic virus responsible for the infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose CSF was analyzed for HSV-1, HSV-2, VZV, EV, EBV, CMV and HHV-6 between 01/01/2014 and 31/12/2024.
* Obtaining informed consent.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include cases from various centers in the Bologna metropolitan area, involving adult and pediatric patients, including newborns, whose CSF was analyzed at the Microbiology Unit of the IRCCS AOUBO, Policlinico di Sant'Orsola, between January 1, 2014, and December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Positivity to different etiological agents (CMV, HSV-1, HSV-2, HHV-6, VZV, EBV, EV) by patient type (pediatric, adult, immunocompetent, immunocompromised) | at enrolment
  For the primary objective, all required molecular investigations of LCRs collected from patients with suspected viral meningitis will be selected from the management software used at the Virology Laboratory between January 1, 2014, and December 31, 2024. Infectious episodes will be identified in relation to the positivity of the viral etiological agent, considering the result (positive or negative) obtained at the time of diagnosis, without having the need to re-examine the sample. An infectious episode is defined as a hospital admission event with a clinical picture of presumed meningitis of viral origin and consequent microbiological confirmation. Therefore, in case of multiple molecular investigations on the same patient during a single hospitalization, it will be considered as the only infectious event. On the other hand, in the event of multiple hospitalizations per single patient with suspected viral meningitis, they will be considered as different infectious episodes.

SECONDARY OUTCOMES:
Clinical course of the patient with episode of viral meningitis, taking into account the type of patient (pediatric, adult, immunocompetent, immunocompromised) and the pathogen | at enrolment
  For secondary objectives, only positive cases of viral etiological agent will be considered and, by accessing the data recorded in the patient's medical record, information regarding symptoms, the outcome of the instrumental examination performed, and the course of the individual hospital stay will be retrieved. Post-discharge, only neurological sequelae will be considered at follow-up at > 6 months, during the follow-up visit with the infectious disease physician.
Distribution of instrumental outcomes of EEC, MRI, CT (normal or non-normal), in the patient with infectious episode, taking into account the patient type (pediatric, adult, immunocompetent, immunocompromised) and the pathogen detected. | at enrolment
  For secondary objectives, only positive cases of viral etiological agent will be considered and, by accessing the data recorded in the patient's medical record, information regarding symptoms, the outcome of the instrumental examination performed, and the course of the individual hospital stay will be retrieved. Post-discharge, only neurological sequelae will be considered at follow-up at > 6 months, during the follow-up visit with the infectious disease physician.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Gabrielli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna; Giulio Virgili, MD, Study Chair — AUSL di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakobsen A, Skov MT, Larsen L, Trier Petersen P, Brandt C, Wiese L, Hansen BR, Luttichau HR, Tetens MM, Helweg-Larsen J, Storgaard M, Nielsen H, Bodilsen J. Herpes Simplex Virus 2 Meningitis in Adults: A Prospective, Nationwide, Population-Based Cohort Study. Clin Infect Dis. 2022 Sep 14;75(5):753-760. doi: 10.1093/cid/ciab1071. Erratum In: Clin Infect Dis. 2022 Nov 30;75(11):2051. doi: 10.1093/cid/ciac790. PMID 34979025
- [Background] Handley G, Pankow S, Bard JD, Yee R, Nigo M, Hasbun R. Distinguishing cytomegalovirus meningoencephalitis from other viral central nervous system infections. J Clin Virol. 2021 Sep;142:104936. doi: 10.1016/j.jcv.2021.104936. Epub 2021 Jul 25. PMID 34352616
- [Background] Aiba Y, Ohshiba S, Horiguchi S, Morioka I, Miyashita K, Kiyota I, Endo G, Takada H, Iwata H. Peripheral hemodynamics evaluated by acceleration plethysmography in workers exposed to lead. Ind Health. 1999 Jan;37(1):3-8. doi: 10.2486/indhealth.37.3. PMID 10052293
- [Background] Lane B, Marks MP, Steinberg GK. Interventional neuroradiology--a new approach to difficult vascular lesions of the brain. West J Med. 1993 Jan;158(1):68-9. No abstract available. PMID 8470393
- [Background] Mazziotti MV, Strasberg SM, Langer JC. Intestinal rotation abnormalities without volvulus: the role of laparoscopy. J Am Coll Surg. 1997 Aug;185(2):172-6. doi: 10.1016/s1072-7515(97)00058-6. PMID 9249085
- See also: Related Info — https://www.amcli.it/documenti/percorsi-diagnostici/
- See also: Related Info — https://www.salute.gov.it/imgs/C_17_eventiEpidemici_2533_comunicato_itemComunicato0_files_itemFiles0_fileAzione.pdf
- See also: Related Info — https://www.salute.gov.it/imgs/C_17_eventiEpidemici_2536_comunicato_itemComunicato0_files_itemFiles0_fileAzione.pdf